CLINICAL TRIAL: NCT01635790
Title: Comparing the Effectiveness and Costs of Bevacizumab to Ranibizumab in Patients With Diabetic Macular Edema (The BRDME Study)
Brief Title: Comparing the Effectiveness and Costs of Bevacizumab to Ranibizumab in Patients With Diabetic Macular Edema (BRDME)
Acronym: BRDME
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. dr. R.O. Schlingemann (Other)
Collaborators: University Medical Center Groningen (Other); Free University Medical Center (Other); Erasmus Medical Center (Other); Radboud University Medical Center (Other); Leiden University Medical Center (Other); UMC Utrecht (Other)
Responsible Party: Sponsor-Investigator, Prof. dr. R.O. Schlingemann, Clinical Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL35860.018.11
Record Dates: First submitted 2012-06-28; First posted 2012-07-10 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Diabetic Macular Edema
Keywords: bevacizumab; ranibizumab; diabetic macular edema; randomized clinical trial
MeSH Terms: interventions — Ranibizumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab (Active Comparator): 0.5 mg ranibizumab. Given as monthly intravitreal injections during 6 months
  Interventions: Drug: Ranibizumab; Drug: Bevacizumab
- Bevacizumab (Active Comparator): 1.25 mg of bevacizumab; Given as monthly intravitreal injections during 6 months
  Interventions: Drug: Ranibizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Ranibizumab — 0.5 mg ranibizumab. Given as monthly intravitreal injections during 6 months
  Other Names: Lucentis
Drug: Bevacizumab — 1.25 mg of bevacizumab; Given as monthly intravitreal injections during 6 months
  Other Names: Avastin

SUMMARY:
The primary objective is to demonstrate the non-inferiority of bevacizumab to ranibizumab in the treatment of patients with DME (OCT central area thickness > 275 μm) as determined by the change in best-corrected visual acuity (BCVA) in the study eye from baseline to month 6.

DETAILED DESCRIPTION:
Objective: To compare the effectiveness and costs of 1.25 mg of bevacizumab to 0.5 mg ranibizumab, given as monthly intravitreal injections during 6 months. It is hypothesized that bevacizumab is non-inferior to ranibizumab regarding its effectiveness.

Study design: This will be a randomized, controlled, double masked, clinical trial in 246 patients in seven academic trial centres in The Netherlands.

Study population: patients 18 years of age or higher with diabetic macular and a best corrected visual acuity BCVA score between 78 and 20 letters in the study eye.

Outcomes: The primary outcome measure will be the change in best-corrected visual acuity (BCVA) in the study eye from Baseline to Month 6.

Secondary outcomes will be amongst others the proportion of patients with a gain of 15 letters or more and/or a BCVA of 20/40 or more at 6 months, and the costs and costs per quality adjusted life-year of the two treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 18 years of age who have signed an informed consent;
2. Patients with Type 1 or Type 2 diabetes mellitus (according to American Diabetes Association or World Health Organization (WHO) guidelines) with glycosylated haemoglobin (HbA1c) less than 12.0% at screening (Visit 1). Patients should be on a dietary, exercise and/or pharmacological program for diabetes. Treatment for diabetes must have been stable for at least 2 months;
3. Patients with visual impairment due to DME (within the EDTRS criteria of clinically significant macular edema) in at least one eye, with a central area thickness >275 ìm, who are eligible for anti-VEGF treatment according to the investigator. If both eyes are eligible, the one with the worse visual acuity, as assessed at visit 1, will be selected by the investigator as the study eye;
4. BCVA equal or more than 24 and less or equal to 78 letters in the study eye at screening using ETDRS- like visual acuity testing charts at a testing distance of 4 meter (approximate Snellen equivalent of 20/32 to 20/320).

Exclusion Criteria:

1. Women of child-bearing potential.
2. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive serum pregnancy test (human chorionic gonadotropin > 5 mIU/ml);
3. Inability to comply with study procedures;
4. Active intraocular inflammation (grade + or above) in either eye at enrolment;
5. Any active infection (e.g., conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) in either eye at the time of enrolment;
6. History of uveitis in either eye at any time;
7. Structural damage within 600 m of the centre of the macula in the study eye likely to preclude improvement in visual acuity following in the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s), epiretinal membrane involving fovea or organized hard exudate plaques;
8. Uncontrolled glaucoma in the study eye at screening (IOP > 24 mmHg on medication or according to investigator's judgment);
9. Neovascularization of the iris in the study eye;
10. Evidence of vitreomacular traction in the study eye;
11. Active untreated proliferative diabetic retinopathy in the study eye;
12. Any intraocular surgery in the study eye within 3 months prior to randomization;
13. History of vitrectomy in study eye regardless of time prior to randomization;
14. Planned medical or surgical intervention during the 6 months study period;
15. Panretinal laser photocoagulation in the study eye within 3 months prior to or during the study;
16. Focal/grid laser photocoagulation in the study eye 3 months prior to study entry;
17. Treatment with anti-angiogenic drugs in the study eye (pegaptanib sodium, anecortave acetate, bevacizumab, ranibizumab, VEGF-Trap, etc.) within 3 months prior to randomization;
18. Use of other investigational drugs at the time of enrolment, or within 3 month or 5 half-lives from enrolment, whichever is longer;
19. History of intravitreal corticosteroids in phakic eye within 18 months prior to randomization or in post-cataract surgery study eye (aphakic or pseudophakic, without damaged posterior capsule) within 4 months prior to randomization;
20. Ocular conditions in the study eye that require chronic concomitant therapy with topical ocular or systemically administered corticosteroids;
21. History of stroke or transient ischemic attack (TIA) within 6 months prior to enrolment;
22. Renal failure requiring dialysis or renal transplant or renal insufficiency with creatinine levels > 2.0 mg/dl at screening;
23. Blood pressure systolic > 165 mm Hg or diastolic > 105 mmHg at screening and randomization;
24. Hypertension or change in antihypertensive treatment within 1 month preceding randomization;
25. Current use of or likely need for systemic medications known to be toxic to the lens, retina or optic nerve, including deferoxamine, chloroquine/hydroxychloroquine (Plaquenil), tamoxifen, phenothiazines and ethambutol;
26. Known hypersensitivity to fluorescein, ranibizumab or bevacizumab or any component thereof or drugs of similar chemical classes;
27. Any type of advanced, severe or unstable disease or its treatment, that may interfere with primary and/or secondary variable evaluations including any medical condition that could be expected to progress, recur, or change to such an extend that it may bias the assessment of the clinical status of the patient to a significant degree or put the patient at special risk;
28. Concomitant conditions in the study eye which would, in the opinion of the investigator, prevent the improvement of visual acuity on study treatment;
29. Ocular disorders in the study eye that may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention during the 6-month study period, including cataract, retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization of any cause (e.g., AMD, ocular histoplasmosis, or pathologic myopia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | 6 months
  Primary outcome measure will be the change in best-corrected visual acuity (BCVA) in the study eye from baseline to month 6.

SECONDARY OUTCOMES:
The proportion of patients with a gain or loss of 15 letters or more | 6 months
  The proportion of patients with a gain or loss of 15 letters or more at 6 months compared to baseline BCVA
Change in leakage on fluorescein angiography | 6 months
  Change in leakage on fluorescein angiography, baseline compared to 6 month exit visit
Change in foveal thickness by optical coherence tomography | 6 months
  The change in foveal thickness (central retinal area) by optical coherence tomography, 6 month exit visit compared to baseline
Number of adverse events | 6 months
  The total number of adverse events that occured during the 6 month study timeframe, with secondary a classification of the types of adverse events
Costs per quality adjusted life-year of the two treatments | 6 months
  The costs per quality adjusted life year of the two treatments, results will be based on the use of standardized health questionnaires (EQ5D or HUI3)
The proportion of patients with a BCVA of 20/40 or more | 6 months
  The proportion of patients with a BCVA of 20/40 or more at 6 months compared to baseline BCVA

CONTACTS AND LOCATIONS:
Overall Officials: Reinier O Schlingemann, MD, PhD, Principal Investigator — Academic Medical Center, Dept. Ophthalmology, Room A2-122, Meibergdreef 9, 1105 AZ Amsterdam, The Netherlands
Locations (1):
- Academic Medical Center, Dept. Ophthalmology,, Amsterdam, Netherlands

REFERENCES:
- [Derived] Fickweiler W, Klaassen I, Vogels IM, Hooymans JM, Wolffenbuttel BH, Los LI, Schlingemann RO; BRDME Research Group. Association of Circulating Markers With Outcome Parameters in the Bevacizumab and Ranibizumab in Diabetic Macular Edema Trial. Invest Ophthalmol Vis Sci. 2016 Nov 1;57(14):6234-6241. doi: 10.1167/iovs.16-20157. PMID 27842163